CLINICAL TRIAL: NCT06842615
Title: Prospective Evaluation of Diagnostic Performance of PanTum Detect Test in Adult Patients With Suspected or Confirmed Macroscopic Solid Pre-malignant or Malignant Lesion(s) Referred to Fludeoxyglucose (18F) PET/CT and in Adult Healthy Population
Acronym: PanTumPET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VEGA 1/0394/24; 2024-514272-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-11; First posted 2025-02-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pre-malignant; Malignant
Keywords: macroscopic; solid lesion; pre-malignant; malignant lesion
MeSH Terms: conditions — Precancerous Conditions

STUDY DESIGN:
Intervention Model Description: PanTum Detect is a multi-tumour screening blood test for the presence of silently growing malignant or pre-malignant lesions.
  PanTum Detect is an Epitope Detection in Monocytes/Macrophages (EDIM) based test technology uses the information contained in the human immune system for detection of pre-malignant or malignant lesions. Higher than normal levels of Apo10 (DNaseX) & transketolase-like protein 1(TKTL1) detected in macrophages of examined individuals gives an indication of potential pre-malignant or malignant lesions.
  The test has an In Vitro Diagnostic (IVD) CE certified specificity of 99% and sensitivity of 97.5%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cancer Group (Experimental): Group A (Patients with suspected or confirmed macroscopic solid pre-malignant or malignant lesion(s) referred to FDG PET/CT): 30 days for patients with confirmed pre-malignant or malignant lesion(s) and 12 months in patients with suspected pre-malignant or malignant lesion(s) for collection of data from routine clinical workup for collection of data for standard of truth.
  Reasons for duration of participation in the study:
  One Pantum detect test is performed in a group of patients with confirmed pre-malignant or malignant lesion(s), at the interval of -30 to 0 or 15-30 days from FDG PET/CT, therefore the duration of inclusion for patients is 1-30 days.
  However, in case of suspected malignancy and negative FDG PET/CT finding, the collection of data from routine clinical follow-up is necessary to confirm or rule-out the presence of macroscopic solid pre-malignant or malignant lesion(s) and establishment of the standard of truth.
  Interventions: Diagnostic Test: Pantum detect test
- Control Group (Other): Reasons for duration of participation in the study: Two Pantum detect test are performed in this group:
  1. first at the inclusion
  2. and the second et the end of 12-month follow-up period
  Reasons for duration of participation in the study:
  When PanTum detect test is performed in this group of participants, the probability of positive finding is low however, to exclude the false negative result the non-detection of macroscopic solid pre-malignant or malignant lesion needs to be confirmed by data from routine clinical follow-up during 12 months. At the end of this follow-up period a second PanTum detect test is performed as a part of clinical follow-up to analyse the concordance of the result over the time. In case of detection of pre-malignant or malignant lesion in healthy before the end of follow-up period, the second Pantum detect test is performed at the time of its diagnosis.
  Therefore, the duration of inclusion for healthy controls is 12 months.
  Interventions: Diagnostic Test: Pantum detect test

INTERVENTIONS:
Diagnostic Test: Pantum detect test — epitope detection in monocyte (EDIM)
  Other Names: FDG PET/CT

SUMMARY:
This prospective phase II trial aims to evaluate the diagnostic performance of multi-cancer epitope diagnosis in monocyte (EDIM) based blood test PanTum detect test for early detection of individuals with pre-malignant or malignant lesion(s).

The intervention in this trial is the PanTum detect test performed in two parallel groups of participants:

Group A:

Adult persons

* with suspected or confirmed macroscopic solid pre-malignant or malignant lesion(s) referred to FDG PET/CT
* meeting the inclusion criteria and not-meeting the exclusion criteria
* Expected number of participants: 67

Group B:

Healthy adult persons

* meeting inclusion criteria meeting the inclusion criteria and not-meeting the exclusion criteria
* Expected number of participants: 67 Control method: uncontrolled

Type of trial: evaluation of diagnostic performance of a diagnostic test with following Primary and Secondary objectives:

Primary Objective

1. To evaluate the sensitivity and specificity of PanTum Detect test in identification of individuals bearing macroscopic solid pre-malignant or malignant lesion(s) Secondary Objectives

1. To evaluate the positive and negative predictive value of PanTum Detect test in identification of individuals bearing macroscopic solid pre-malignant or malignant lesion(s)
2. To assess the concordance of result of PanTum Detect test with result of FDG PET/CT for macroscopic solid pre-malignant or malignant lesion(s)
3. To analyse the most frequent causes of false results of PanTum Detect test
4. To analyze the concordance rate of PanTum Detect test No1 and No2
5. To refine the interpretation criteria of PanTum Detect test
6. To analyse the subject´s willingness to participate on the trial
7. To analyse the subject´s experience with participation on the trial

DETAILED DESCRIPTION:
PanTum Detect is a multi-tumour screening blood test for the presence of silently growing malignant or pre-malignant lesions.

PanTum Detect is an Epitope Detection in Monocytes/Macrophages (EDIM) based test technology uses the information contained in the human immune system for detection of pre-malignant or malignant lesions. Higher than normal levels of Apo10 (DNaseX) & transketolase-like protein 1(TKTL1) detected in macrophages of examined individuals gives an indication of potential pre-malignant or malignant lesions.

23 The test has an In Vitro Diagnostic (IVD) CE certified specificity of 99% and sensitivity of 97.5%.

For details on Intervention please refer to Appenidix 13.1 Manual-Test Kit Booklet - IFU_V04-TB-ZE-EN_DE-V4.0

In this trial, PanTum detect test is performed in two groups of participants:

In Group A of included participants:

In participants with confirmed pre-malignant or malignant lesion(s) the PanTum test is performed at the time of inclusion and its diagnostic performance will be assessed in comparison with standard of truth for fulfilment of the primary objective.

In participants with suspected pre-malignant or malignant lesion(s) the PanTum test is performed at the time of inclusion and at the end of follow-up period of 12 months and its diagnostic performance will be assessed in comparison with standard of truth for fulfilment of the primary and secondary objective. The result of PanTum Detect test performed at the end of the follow-up period will be used for fulfilment of secondary objective.

In Group B of included participants:

In healthy asymptomatic individuals at the time of inclusion and at the end of 12-month follow-up period. Its diagnostic performance at inclusion will be assessed in comparison with standard of truth.

The result of PanTum detect test at the end of follow-up period will be used for fulfilment of secondary objective.

Total duration of trial intervention for each participant is as follows:

Group A (Patients with suspected or confirmed macroscopic solid pre-malignant or malignant lesion(s) referred to FDG PET/CT): 30 days for patients with confirmed pre-malignant or malignant lesion(s) and 12 months in patients with suspected pre-malignant or malignant lesion(s) for collection of data from routine clinical workup for collection of data for standard of truth.

Reasons for duration of participation in the study:

One Pantum detect test is performed in a group of patients with confirmed pre-malignant or malignant lesion(s), at the interval of 0-30 days from FDG PET/CT, therefore the duration of inclusion for patients is 1-30 days.

However, in case of suspected malignancy and negative FDG PET/CT finding, the collection of data from routine clinical follow-up is necessary to confirm or rule-out the presence of macroscopic solid pre-malignant or malignant lesion(s) and establishment of the standard of truth.

In this group of individuals, the second PanTum detect test may be performed at the end of follow-up period to analyze the concordance of result of PanTum detect test over the time Therefore, the participation of all subjects in the study is set-up to 12 months.

Group B (Adult healthy individuals): 12 months

Reasons for duration of participation in the study: Two Pantum detect test are performed in this group:

3. one at the inclusion 24 4. and the second et the end of 12-month follow-up period

Reasons for duration of participation in the study:

When PanTum detect test is performed in this group of participants, the probability of positive finding is low however, to exclude the false negative result the non-detection of macroscopic solid pre-malignant or malignant lesion needs to be confirmed by data from routine clinical follow-up during 12 months. At the end of this follow-up period a second PanTum detect test is performed as a part of clinical follow-up to analyse the concordance of the result over the time. In case of detection of pre-malignant or malignant lesion in healthy before the end of follow-up period, the second Pantum detect test is performed at the time of its diagnosis.

Therefore, the duration of inclusion for healthy controls is 12 months.

Randomization:

The trial intervention is performed in Group A and Group B per inclusion criteria.

The blinding described below may be considered as a surrogate randomization. No other forms of randomization are applicable in this trial.

Blinding:

* The laboratory performing the Pantum detect test is blinded to clinical context of the participant with corresponding blood sample.
* The independent assessor is blinded to result of PanTum detect test for establishment of the standard of truth No within-trial transition is possible in tris trial As this is the trial with diagnostic test the dose escalation or dose-ranging is not applicable.

Method of Assignment to Trial Intervention: all included participant will receive the same intervention, as per protocol This is a single centre trial.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet all the following criteria:

Group A

* Age 18-88 years at inclusion (Man, Woman)
* Suspected or confirmed macroscopic solid pre-malignant or malignant lesion(s)
* Availability of result of FDG PET/CT performed -30 to-15 days or up to +30 days from trial intervention and performed as a standard of care
* Willingness to undergo trial intervention
* Signed informed consent
* Absence of any of exclusion criteria Group B
* Age 18-88 years at inclusion (Man, Woman)
* Considered as free of pre-malignant or malignant lesion(s) at the time of inclusion
* Willingness to undergo trial intervention
* Signed informed consent
* Absence of any of exclusion criteria

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this trial: For Group A and B

1. Acute Illness, Organ Transplantation, Surgeries, and injuries are an exclusion criteria: e.g. bone fracture, deep cut (deeper 0.5 cm and/or larger than 1 cm), abrasion (greater than 5 cm in diameter), open wound, contusion, torn ligaments, blood in the stool, blood in the urine. After successful recovery the waiting period must be 8 weeks.
2. Medication: Any treatment or activity that could impact the immune system must be considered as an exclusion criteria.These includes.

   1. Steroid-, chemo-, radio therapy in last 8 weeks
   2. Immunesuppression using following active ingredients; Methotrexate, Cyclosporine, Azathioprine, Tacrolimus, Mycophenolate, Rapamycin, Sirolimus, Mycophenolat-Mofetil in last 8 weeks.
   3. Granulocyte-Macrophage Colony-Stimulating Factor (GM-SCF); Molgramostim, Sargramostim in last 8 weeks o Amygdalin (Vitamin B17) in last 4 weeks
   4. Immune modulation using Corticosteroids, Glucocorticoids and Colchicine (Cortison/hydrocortisone >5 mg/day, Budesonid >5 mg/day) in last 4 weeks
   5. Non-Steroidal anti-inflammatory drugs (NSAIDs) & CGRP including in last 2 weeks. An occasional use of Ibuprofen, Paracetamol and Aspirin is not an exclusion criteria.
   6. Antibiotics and Antifungals in last 2 weeks
3. Vaccination: any vaccination in last 4 weeks.
4. Infection: Acute Bacterial, Viral infection and Fungal infection in last 2 weeks.
5. Imaging Investigation using contrast medium in last 2 weeks.
6. Dialysis on the day of blood draw.
7. Genetic disorder such as thrombocytopenia may leads to rejection of test due to reduced amount of Blood Cells.

For Group B only:

1. Previous and Current Cancer: In case of previously diagnosed and successfully treated Tumour & cancer, the PanTum Detect test should be done 5 years after the successful treatment & cure. This applies to all kind of Tumour and Cancers. all currently ongoing cancer treatments and newly diagnosed cancer including ongoing diagnostic procedures are an exclusion criterion

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-05-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
PanTum test | 1st day
  To evaluate the sensitivity and specificity of PanTum Detect test in identification of individuals bearing macroscopic solid pre-malignant or malignant lesion(s) Localization of macroscopic solid pre-malignant or malignant lesion(s)

SECONDARY OUTCOMES:
positive and negative predictive value of PanTum Detect test | 1st day
  To evaluate the positive and negative predictive value of PanTum Detect test in identification of individuals bearing macroscopic solid pre-malignant or malignant lesion(s)
concordance of result of PanTum Detect test | 1st day
  To assess the concordance of result of PanTum Detect test with result of FDG PET/CT for macroscopic solid pre-malignant or malignant lesion(s) Discordant result of PanTum Detect test and the result of FDG PET/CT for macroscopic solid pre-malignant or malignant lesion(s)
false results of PanTum Detect test | 1st day
  To analyse the most frequent causes of false results of PanTum Detect test
concordance rate of PanTum Detect test | 12th month
  To analyse the concordance rate of PanTum Detect test No1 and No2 Concordant result of PanTum Detect test No1 and No2

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No